CLINICAL TRIAL: NCT03700437
Title: Randomized Controlled Pilot Study to Evaluate Fasting-mimicking Diet in Patients Receiving Chemo-immunotherapy for Treatment of Metastatic Non-small Cell Lung Cancer
Brief Title: Fasting-mimicking Diet With Chemo-immunotherapy in Non-small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Shadia Jalal, Associate Professor of Clinical Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IUSCC-0662
Record Dates: First submitted 2018-09-25; First posted 2018-10-09 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: fasting; diet; chemo-immunotherapy; lung cancer; circulating tumor cells
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Fasting; Lung Neoplasms; Neoplastic Cells, Circulating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fasting-Mimicking Diet (FMD) (Experimental): Participants randomized to the intervention arm (FMD) will be provided with Chemolieve®, a plant-based FMD that provides ~300 calories/fasting day and includes all the food to be consumed during the dietary intervention including supplements
  Subjects will start the diet 3 days prior to chemo-immunotherapy and continue on the first day of chemo-immunotherapy for the first 4 cycles of therapy.
  Interventions: Other: Fasting-Mimicking Diet

INTERVENTIONS:
Other: Fasting-Mimicking Diet — Chemo-immunotherapy + FMD (fast-mimicking diet)

SUMMARY:
The purpose of this study is to learn the effects of fasting on cancer cells while you get maintenance treatment.

DETAILED DESCRIPTION:
Cancer cells use an increased supply of glucose to make energy and do not have protection against fasting that normal cells do. Because of this, researchers would like to study how fasting may help chemotherapy target cancer cells instead of normal cells. Initial studies suggest that fasting may decrease the side effects of chemotherapy and increase the chances of your cancer responding to the chemotherapy. Patient populations will have non-small cell lung cancer in which chemo-immunotherapy with carboplatin/pemetrexed and pembrolizumab have been recommended to treat the cancer as part of standard care.

Primary Objective 1. To determine the feasibility and compliance of administering a fasting-mimicking diet (FMD) in patients with advanced NSCLC receiving maintenance therapy

Secondary Objectives

1. To assess a patient's willingness to fast for second cycle

Correlative Objectives

1. To assess DNA damage via measurement of γ-Η2ΑΧ foci in PBMCs at baseline and following one cycle of FMD (day 21 or day 28)
2. To assess spheroid formation from circulating tumor cells (CTCs) isolated from patients post FMD as compared to baseline (prior to fasting)
3. To measure the changes in immune markers prior to and after administering the FMD

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years at the time of informed consent
2. Ability to provide written informed consent and HIPAA authorization
3. Eastern cooperative group (ECOG) performance status of 0 to 2
4. Histologically confirmed Non-Small Cell Lung Cancer (NSCLC) and have advanced disease.
5. BMI ≥ 19
6. Patients should be on maintenance therapy for advanced NSCLC as defined as treatment with single agent immunotherapy, single agent chemotherapy plus immunotherapy or single agent molecularly targeted therapy for a minimum of 2 months prior to study entry
7. If a patient is on a treatment that lowers their ANC, their ANC has to be ≥ 1500 on the first day of fasting

Exclusion Criteria:

1. Self-reported weight loss of > 10% in the 6 weeks prior to study entry
2. History of diabetes mellitus or patients with a known recent elevated A1c > 6
3. History of symptomatic hypoglycemia
4. Prior therapies with inhibitors of IGF-1 such as

   1. Linsitinib
   2. Picropodophyllin
5. Concurrent use of somatostatin
6. Concurrent use of immunosuppressive medications including sirolimus, tacrolimus, mycophenolate mofetil, azathioprine, prednisone, dexamethasone, or cyclosporine
7. Significant food allergies (screening checklist in Appendix 3) which would make the subject unable to consume the food provided
8. History or current evidence of any medical or psychiatric condition, therapy that may confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the participating subject as deemed by the treating investigator.
9. Pregnant or lactating females are not eligible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-02 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Proportion of the patients who can finish the FMD without serious adverse events | Between screening/baseline (28 to 4 days before Cycle 1 Day 1) and Cycle 1 Day 21 or 28 (Cylces last 21 or 28 days, based on treatment)
  To assess feasibility, compliance will be measured by a daily log

CONTACTS AND LOCATIONS:
Overall Officials: Shadia Jalal, MD, Principal Investigator — Indiana University
Locations (3):
- United States (3):
  - Eskenazi Hospital, Indianapolis, Indiana
  - Indiana University Hospital, Indianapolis, Indiana
  - Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No